CLINICAL TRIAL: NCT01004575
Title: Clinical Evaluation of Kaname Cobalt-Chromium Coronary Stent System in the Treatment of Patients With Coronary Artery Disease
Brief Title: Safety and Efficacy Study of Kaname Coronary Stent System for the Treatment of Patients With Coronary Artery Disease
Acronym: KARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T111E4
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Coronary Artery Disease; Angioplasty, Transluminal, Percutaneous Coronary
Keywords: stents; bare metal stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kaname (Experimental): patients that are treated by implanting Kaname Cobalt-Chromium coronary stent
  Interventions: Device: implantation of Kaname Cobalt-Chromium coronary stent

INTERVENTIONS:
Device: implantation of Kaname Cobalt-Chromium coronary stent — implantation of Kaname Cobalt-Chromium coronary stent
  Other Names: Kaname; Cobalt-chromium; coronary stent

SUMMARY:
The purpose of this study is to assess whether the new Kaname coronary stent is safe and effective for the treatment of patients with coronary artery disease.

DETAILED DESCRIPTION:
Current treatments for coronary artery disease include conservative treatment (drug therapies) and invasive techniques that help increase blood flow to ischemic or oxygen-deprived regions of the heart. Among the invasive techniques the most frequently used are coronary artery bypass graft surgery (CABG), and percutaneous transluminal coronary angioplasty (PTCA) without or with stents (bare metal stents (BMS) or drug eluting stents (DES)) implantation. However, all of those treatments have limitations and their effectiveness is diminished under certain circumstances. Therefore, it is essential to tailor therapy for each individual patient considering the overall patient's condition, disease severity and progression as well as concomitant diseases. The question of selection of appropriate stent for each individual patient is still unresolved and most of the physicians either follow international or national guidelines or scientific wisdom.

Although the efficacy of DES is undisputable in restenosis prevention, because some patients could have adverse outcomes from a DES, they should be used selectively in those who are most likely to benefit, and in that decision process several important issues should be addressed such as:Patients' adherence to post-stenting therapy, Bleeding risk, Need for elective surgery, Risk for restenosis, Risk for stent thrombosis. It is still believed that many patients will do well with BMSs and that this technology requires further refinements to improve outcome. For the above reasons Terumo has designed the new coronary BMS, Kaname™, a balloon expandable Cobalt-Chromium (CoCr) stent pre-mounted onto a high pressure, semi-compliant balloon on a rapid exchange delivery catheter. The Kaname stent is the subject of the current prospective, multi-centre KARE study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old.
* Patient is eligible for PCI and acceptable candidate for CABG.
* Clinical evidence of ischemic heart disease and/or a positive functional study. Documented stable angina pectoris (CCS 1, 2, 3 or 4) or unstable angina pectoris with documented ischemia (Braunwald Class IB-C, IIB-C, or IIIB-C), or documented silent ischemia.
* The target lesion or target vessel meets all the following criteria;a) is a single de novo lesion or restenotic post-PTCA (non-stented) lesion in one native coronary artery.b)The stenosis of target lesion is ≥ 50% and < 100% c)The target lesion length must be ≤ 25 mm d)The target reference vessel diameter must be suitable for treatment with stents between 2.5 and 4.0 mm long
* Patient has been informed of the nature of the study, understands the study requirements and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee of the respective clinical site.
* The patient is able to comply with all specified follow-up evaluations.

Exclusion Criteria:

* Most recent LVEF of the patient is < 25%.
* Known allergies to the following: aspirin, Clopidogrel bisulfate, Prasugrel or Ticlopidine, heparin, cobalt, chromium, nickel, or contrast agent (that cannot be adequately premedicated).
* A platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
* WBC count < 3500 cells/mm3.
* Evidence of MI with positive Troponin within 72 hours of the intended treatment.
* Previous PCI (<30 days) anywhere within the target vessel.
* Planned interventional treatment of any non-target vessel <30 days post-procedure will be required. Planned intervention on the target vessel or on a significant lesion of > 50% stenosis anywhere within the target vessel after the index procedure will be required.
* The target lesion requires treatment with a device other than PTCA balloon prior to stent placement. (e.g. but not limited to directional coronary atherectomy, excimer laser, rotational atherectomy, etc.).
* Previous stenting anywhere within the target vessel.
* Target vessel has evidence of thrombus.
* Excessive tortuousity (> 60°) of the target vessel proximal to the target lesion (visual estimate).
* Either of the following characteristics in the target lesion (visual estimate): a)Ostial target lesion or bifurcation lesion b)Target lesion involves a side branch > 2mm in diameter c) Target lesion has excessive tortuousity (> 45°)d)Moderate to severely calcified lesion which can not be successfully predilated e)Target lesion is located in or supplied by an arterial or venous bypass graft f)Significant (> 40%) stenosis proximal or distal to the target lesion. g) A complete occlusion (TIMI flow 0 or 1).
* Target lesion located in left main trunk.
* Stroke or transient ischemic attack < prior 180 days.
* Active peptic ulcer or upper GI bleeding < prior 180 days.
* The patient has bleeding hemorrhagic diathesis or coagulopathy. The patient will refuse a blood transfusion.
* The patient has a widespread peripheral vascular disease.
* Acute or chronic renal dysfunction (creatinine > 2.0 mg/dl).
* The patient requires multiple stent implantations for a tandem lesion.
* Life expectancy < 1 year.
* Patient is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints. Note: Trials requiring extended follow-up for products that were investigational, but have become commercially available since then, are not considered investigational trials.
* In the investigators opinion patient has a co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study.
* Patient is in cardiogenic shock.
* Female of child-bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Freedom from Target vessel failure TVF | 6 months post-procedure
  Freedom from Target vessel failure TVF defined as composite of clinically driven target vessel revascularization (TVR)myocardial infarction or cardiac death that could not be clearly attributed to a vessel other than the target vessel.

SECONDARY OUTCOMES:
Freedom from TVF for patients treated with ≥ 3 mm stents. | 6 months post-procedure
  Freedom from Target Vessel Failure (composite of clinically driven TVR, myocardial infarction or cardiac death that could not be clearly attributed to a vessel other than the target vessel) for patients treated with ≥ 3 mm stents.
Freedom from TVF for patients treated with 2.5 and 2.75 mm stents | 6 months post-procedure
  Freedom from Target Vessel Failure (composite of clinically driven TVR, myocardial infarction or cardiac death that could not be clearly attributed to a vessel other than the target vessel) for patients treated with 2.5 and 2.75 mm stents
Freedom from TVF | 30 days,12 months and 3 and 5 years post-procedure
  Freedom from Target Vessel Failure (composite of clinically driven TVR, myocardial infarction or cardiac death that could not be clearly attributed to a vessel other than the target vessel)
Clinically driven target lesion revascularization (TLR) free rate . | 30 days, 6 and 12 months, 3 and 5 years post-procedure
  Clinically driven target lesion revascularization (TLR) free rate
Clinically driven target vessel revascularization (TVR) free rate. | 30 days, 6 and 12 months, 3 and 5 years post-procedure
  Clinically driven target vessel revascularization (TVR) free rate.
Device success | Baseline procedure
  Device success defined as achievement of a residual diameter stenosis of < 50% by QCA or < 30% by visual estimate, using the assigned device only.
Lesion success | Baseline procedure
  Lesion success defined as the attainment of residual diameter stenosis of < 50% by QCA or < 30% by visual estimate, using any percutaneous method.
Procedure success | During baseline hospital stay
  Procedure success defined as achievement of a final diameter stenosis of < 50% by QCA or < 30% by visual estimate, using any percutaneous method, without MACE (composite of cardiac death, MI and TLR) .
Angiographic in-stent acute gain | Baseline procedure
  Angiographic in-stent acute gain at the end of the procedure
Angiographic in-stent and in-segment binary restenosis rate (≥ 50%) diameter stenosis | 6 months post-procedure
  Angiographic in-stent and in-segment binary restenosis rate (≥ 50%) diameter stenosis
Angiographic in-stent, in-segment, proximal, and distal minimum lumen diameter (MLD) | 6 months post-procedure
  Angiographic in-stent, in-segment, proximal, and distal minimum lumen diameter (MLD)
In-stent late-loss | 6 months post-procedure
  In-stent late-loss (as measured by QCA) defined as the difference between the post-procedure minimal lumen diameter (MLD) and the follow-up MLD.
% Diameter Stenosis, in-stent and in-segment . | 6 months post-procedure
  % Diameter Stenosis, in-stent and in-segment.
Neointimal hyperplasia volume as measured by intravascular ultrasound. | 6 months post-procedure
  Neointimal hyperplasia volume as measured by intravascular ultrasound at 6 months post-procedure
Major adverse cardiac events (MACEs) rate . | 30 days, 6 and 12 months, 3 and 5 years post-procedure
  Major adverse cardiac events (MACEs: composite of cardiac death,, myocardial infarction and TLR) rate.
Serious adverse event rate . | 30 days, 6 and 12 months, 3 and 5 years post-procedure
  Serious adverse event rate.
Device failure . | Baseline procedure
  Any device failure

CONTACTS AND LOCATIONS:
Overall Officials: Didier Carrie, Prof Dr, Principal Investigator — CHU Rangeuil, 31059 Toulouse, France
Locations (17):
- France (5):
  - Hopital Cardiovasculaire et Pneumologie Louis Pradel, Lyon
  - CHU NORD, Nantes
  - Clinique les Franciscaines, Nîmes
  - Hopital d'Instructions des Armées du Val de Grace, Paris
  - CHU Rangeuil, Toulouse
- Germany (3):
  - Klinikum Fulda gAG, Fulda
  - Klinikum Ludwigshafen, Ludwigshafen
  - Klinikum des Johannes Gutenberg Universität, Mainz
- Italy (3):
  - Ospedale Careggi, Florence
  - Policlinico Milano, Milan
  - Ospedale Civico Palermo, Palermo
- Serbia (3):
  - Clinical Centre of serbia, Belgrade
  - Clinical Hospital Center Zemun, Belgrade
  - Institute for Cardiovascular Disease Dedinje, Belgrade
- Spain (3):
  - Hospital Clinico San Carlos, Madrid
  - Hospital La Paz, Madrid
  - Hospital Meixoeiro, Vigo